CLINICAL TRIAL: NCT01163136
Title: Decision Making in Serious Pediatric Illness
Acronym: DSPI
Status: Completed | Type: Observational
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Other Study IDs: 10-007447; 1R01NR012026-01 (NIH)
Record Dates: First submitted 2010-07-13; First posted 2010-07-15 (Estimated); Last update posted 2017-10-03 (Actual); Status verified 2017-09

CONDITIONS: Parental Decision Making for Seriously Ill Children
Keywords: Parental decision making; Decision Making in Serious Pediatric Illness (DSPI); palliative care decision making

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study will look at a cohort of parents whose children are confronting life-threatening illnesses in intensive care, palliative care, and complex care settings, to test whether parents with higher levels of hopeful patterns of thinking are subsequently more likely a) to change the "level of care" order status of their child (as an important and demonstrable example of adapting goals); b) to reprioritize goals for the child when they are reassessed regarding goals ; and c) to report a higher degree of achieving self-defined 'good parent' attributes.

DETAILED DESCRIPTION:
Parents making medical decisions for a child living with a life-threatening condition confront, sometimes repeatedly, an extremely daunting task: how to decide when to set aside the therapeutic goal of cure or of life prolongation and instead prioritize the goals of comfort or quality of life.

This study will look at a cohort of parents whose children are confronting life-threatening illnesses in intensive care, palliative care, and complex care settings, to test whether parents with higher levels of hopeful patterns of thinking are subsequently more likely a) to change the "level of care" order status of their child (as an important and demonstrable example of adapting goals); b) to reprioritize goals for the child when they are reassessed regarding goals ; and c) to report a higher degree of achieving self-defined 'good parent' attributes.

We hypothesize that parents with higher levels of hopeful patterns of thinking subsequently will be:

More likely to enact a limit of intervention order. More likely, upon explicit formal reassessment, to reprioritize goals for the child.

More likely to report a higher degree of achieving self-defined 'good parent' attributes.

ELIGIBILITY:
Inclusion Criteria:

* Parents of children who are patients at The Children's Hospital of Philadelphia (CHOP) admitted to the neonatal, pediatric, or cardiac intensive care unit (NICU, PICU, or CICU), or who have been referred to the Pediatric Advanced Care Team (PACT) for palliative care services. A patient is eligible when the patient's attending physician considers it likely that parents will have major treatment decisions to make for their child within the coming 12 to 24 months.

Exclusion Criteria:

* Non English-speaking parents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Parents of children of age < 18 years or cognitively impaired such that their parents make all medical decisions on their behalf; and of either gender and any race/ethnicity who are patients at The Children's Hospital of Philadelphia (CHOP) admitted to the neonatal, pediatric, or cardiac intensive care unit (CICU), neonatal intensive care unit (NICU), or pediatric intensive care unit (PICU), or who have been referred to the Pediatric Advanced Care Team (PACT) for palliative care services.
Sampling Method: Non-Probability Sample
Enrollment: 358 (Actual)
Dates: Start 2010-07; Primary Completion 2014-11 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Parents' reprioritized goals | up to 2 years
  Parents, when interviewed every 4 months for up to 2 years, are asked what the goals of care are for their child, and if the priority of those goals has changed.

SECONDARY OUTCOMES:
Parents' self-defined 'good parent' attributes | up to 2 years
  Parents, when interviewed every 4 months for up to 2 years, are asked how they assess their achievement of attributes of being a good parent to their ill child

CONTACTS AND LOCATIONS:
Overall Officials: Chris Feudtner, MD, PhD, MPH, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States